CLINICAL TRIAL: NCT06834555
Title: Can Mobile Phone Thermal Imaging Provide an Ambulatory Assessment of Incompetent Perforator Veins?
Brief Title: Mobile Phone Thermal Imaging Assessment of Incompetent Perforator Veins
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Second Provincial General Hospital (Other)
Responsible Party: Principal Investigator, Hao Liu, Attending Doctor, Guangdong Second Provincial General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-KY-KZ-432
Record Dates: First submitted 2025-02-08; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Chronic Venous Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- insufficient perforated veins in CVD patients (Experimental): The patient was supine, and the lower limb was naturally relaxed on a 20cm high stent to drain blood from the vein. The leg temperature was lowered with a cold towel at 2-6 ° C for five minutes. A tourniquet was applied to the upper 1/3 of the thigh and the level of the fibula of the lower leg with enough pressure to block the great saphenous vein and the small saphenous vein. The patient is then asked to stand. The smart phone and the supporting thermal imaging system were used to conduct continuous real-time imaging and take photos of the front, bilateral and rear of the thigh and lower leg. The hot spot of "rapid rewarming" of the lower limb was marked with a marker.
  Interventions: Diagnostic Test: Mobile phone thermal imaging

INTERVENTIONS:
Diagnostic Test: Mobile phone thermal imaging — The patient was supine, and the lower limb was naturally relaxed on a 20cm high stent to drain blood from the vein. The leg temperature was lowered with a cold towel at 2-6 ° C for five minutes. A tourniquet was applied to the upper 1/3 of the thigh and the level of the fibula of the lower leg with enough pressure to block the great saphenous vein and the small saphenous vein. The patient is then asked to stand. The smart phone and the supporting thermal imaging system were used to conduct continuous real-time imaging and take photos of the front, bilateral and rear of the thigh and lower leg. The hot spot of "rapid rewarming" of the lower limb was marked with a marker.

SUMMARY:
Chronic venous disease is a common disease of the lower limbs. Severe CVD can lead to lower limb swelling, pigmentation, and repeated skin ulceration, which seriously affects patients' quality of life. About 10.5% to 92.7% of CVD patients with recurrent varicose veins had insufficient perforating veins. Treatment of these IPVs can promote venous ulcer healing and reduce the recurrence rate of venous ulcers. Accurate assessment and positioning of insufficient perforating veins in the lower leg is a key step in developing a personalized treatment strategy. At present, Color Doppler ultrasonography performed in the upright position in combination with the Valsalva maneuver or local pressure of the limb is regarded as the "gold standard" for the diagnosis of perforating veins insufficiency. However, in China, a large number of perforating veins insufficiency are diagnosed by venography. Because the majority of Chinese vascular surgeons are not versatile in vascular ultrasound examination and venous ultrasound protocols vary from institution to institution. A non-functioning valve in an insufficient perforated vein allows blood to flow retrograde from a deep vein to a superficial vein. Some researchers have shown that the venous blood temperature of deep veins is higher than that of superficial veins. Thus, the retrograde flow of "warm blood" from the deep vein to the superficial vein increases the skin temperature located on the insufficient perforated vein. This study tested the feasibility of a smartphone and its compatible portable thermal imaging device as a tool for assessing insufficient perforated vein. The objective is to study the sensitivity and specificity of smartphone thermal imaging in diagnosing and locating the insufficient perforated vein in CVD patients.

ELIGIBILITY:
Inclusion Criteria:

A diagnosis of CVD by vascular surgeon, classified C0 to C6 according to CEAP (Clinical-Etiology - Anatomy - Pathophysiology) No history of lower extremity surgery The body mass index (BMI) is 18 to 35 kg/m2

Exclusion Criteria:

deep vein thrombosis heart disease peripheral artery disease chronic liver disease chronic kidney disease pregnancy severe obesity (BMI ≥35 kg/m2)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity of smartphone thermal imaging in diagnosing and locating the insufficient perforated vein in CVD patients | 10 months

IPD SHARING:
Plan to Share IPD: No